CLINICAL TRIAL: NCT03763825
Title: A Pilot Trial of the Mini-AFTERc Intervention to Manage Fear of Cancer Recurrence in Breast Cancer Patients
Brief Title: Mini-AFTERc Intervention for Fear of Cancer Recurrence
Acronym: Mini-AFTERc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of St Andrews (Other)
Collaborators: University of Stirling (Other); University of Surrey (Other); Swansea University (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Prof G Humphris, Professor of Health Psychology, University of St Andrews
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 249571
Record Dates: First submitted 2018-10-23; First posted 2018-12-04 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Fear of Cancer
Keywords: fear of recurrence; cancer; brief intervention; telephone counselling; following primary cancer treatment
MeSH Terms: conditions — Breast Neoplasms; Pathophobia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patient will receive the Mini-AFTERc intervention after completion of primary breast cancer treatment.
  Interventions: Behavioral: Mini-AFTERc
- Control group (No Intervention): Patients will receive usual care after completion of primary breast cancer treatment.

INTERVENTIONS:
Behavioral: Mini-AFTERc — Structured 30-45 minute telephone discussion based on health psychology theory and CBT principles.
  Arms: Intervention group

SUMMARY:
People treated for breast cancer often live with an ongoing fear that the cancer will recur. This fear may develop and impact on their mental health and quality of life. The Mini-AFTERc study is a pilot trial of a brief cognitive behavioural communication intervention, designed to reduce fear of cancer recurrence (FCR) in breast cancer patients. This pilot trial aims to determine the acceptability and practicality of introducing the Mini-AFTERc intervention into everyday practice, and inform the development of a full randomised controlled trial.

DETAILED DESCRIPTION:
The objectives of this pilot trial are as follows:

1. To develop a procedure for training breast cancer nurses (BCN) in the delivery of the Mini-AFTERc intervention and introduce the intervention into current NHS service provision for breast cancer patients.
2. To collect data to pilot and test recruitment (of breast cancer nurses and breast cancer patients), the fidelity of intervention elements, the acceptability to participants (primary and secondary outcomes) and detailed economic indicators for a full trial.
3. Apply a formal decision making framework (ADePT) to determine a profile of factors to reveal potential difficulties and appraise solutions prior to a full trial.

This study is a multicentre controlled pilot trial of the Mini-AFTERc intervention and will take place in 4 breast cancer centres in NHS Scotland health boards, including Fife, Highlands, Lothian and Tayside. Two centres will deliver the intervention (Fife and Lothian) and 2 centres will deliver usual care to patients, acting as control centres (Highlands and Tayside). The project will be delivered in 3 phases:

Phase 1 will include the development and delivery of the Mini-AFTERc intervention training package for breast cancer nurses.

Phase 2 will include patient recruitment and data collection. There will be 2 intervention centres and 2 control centres across NHS Scotland. Patients who have completed their primary breast cancer treatment, will be screened for moderate FCR (scoring ≥10 and <15 on the Fear of Cancer Recurrence 4-item Scale; FCR4). Breast cancer nurses will deliver the intervention by telephone in intervention centres, which will be audio recorded. Patients will complete a satisfaction questionnaire after the intervention (CARE and MISS). Follow-up questionnaires measuring fear of cancer recurrence, anxiety and depression and quality of life outcomes (FCR4, HADS, EQ-5D) will be delivered via a smartphone app at 2 weeks, 1 month and 3 months following intervention or 3 weeks, 5 weeks and 13 weeks following screening for the control group. Semi-structured interviews with 20% of patients and all nurses will be conducted to assess experiences and acceptability of the intervention.

Phase 3 will conduct data analysis and trial evaluation. Screening and follow-up data will be quantitatively analysed, including structured equation modelling. Interviews will be subject to framework analysis based on normalisation process theory (NPT). The pilot trial will be systematically evaluated using a process of decision making after pilot and feasibility trials (ADePT).

The findings will help to understand if this brief intervention can be implemented in everyday practice and can reduce FCR. They will also inform the practicality of implementation of a larger-scale randomised trial.

ELIGIBILITY:
Patient inclusion criteria for screening:

* Completed primary cancer treatment.
* Cancer-free.
* Female.
* Responsible clinician agrees to their participation.

Patient inclusion criteria for trial:

* Score 'moderate' (≥10 and <15) on the Fear of Cancer Recurrence 4-item scale (FCR4) during screening.

Patient exclusion criteria:

* Not completed primary cancer treatment.
* Not cancer-free.
* Male.
* A diagnosed psychotic disorder, known to the cancer service, for which the patient is currently receiving treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2019-06-13 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with nurse communication during the Mini-AFTERc intervention | 1 week post intervention
  Assessed using the Consultation and Relational Empathy (CARE) measure, validated for use in secondary care (Mercer et al. 2004). The CARE measure asks patient to rate their nurses' communication skills on 10 communication and empathy domains (e.g. 'How was your nurse at fully understanding your concerns?'). Patients rate nurses from 1 ('Poor') to 5 ('Excellent') for each of the 10 domains.

SECONDARY OUTCOMES:
Fear of cancer recurrence level - FCR4 | 3 months
  The FCR4 is a 4-item measure designed to assess patient anxiety, worry and strong feelings associated with the return of cancer (e.g. 'I am afraid that my cancer may recur'). The research group has validated the FCR4 as an accurate measure of cancer recurrence fears in breast cancer patients that is fit for routine use in clinical services (Humphris, Watson, Sharpe, & Ozakinci, 2018). Each question in the FCR4 is rated by the patient on a scale of 1 ('Not at all') to 5 ('All the time'). A cumulative score of ≥10 (60 Percentile) across all 4 items is defined as 'moderate' fear of cancer recurrence and a cumulative score of ≥15 is defined as 'high' fear of cancer recurrence.
Depression and anxiety symptoms - Hospital Anxiety and Depression Scale (HADS) | 3 months
  The HADS is a 14-item assessment tool used to screen for anxiety and depression the general medical population (Zigmond & Snaith, 1983). The HADS is well established tool and has been employed in a multitude of medical settings, including oncology, to assess patients' mental health (Hartung et al., 2017; Vodermaier & Millman, 2011). The HADS assesses two domains, depressionand anxiety. Patients report symptoms of depression and anxiety in the last week on a 4-point Likert scale, from 0 (e.g. "Not at all") to 3 (e.g. "Most of the time").
Health-related quality of life - EuroQol 5 Dimension Measure of Quality of Life (EQ-5D) | 3 months
  The EQ-5D is a standardised instrument of health-related quality of life, developed by the EuroQol Group (Herdman et al., 2011). The EQ-5D assesses 5 dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D contains 6-items, 5 of these items assess each of the 5 dimensions and are rated on a 5-level (5L) scale. The final item is a measure of health state, which is rated on a scale of 0 ('worst imaginable health state') to 100 (Best imaginable health state').
Nurses' perceived acceptability of the Mini-AFTERc intervention as part of routine cancer care - Determined by theory driven semi-structured interviews | Within 1 month of delivering final intervention
  Semi-structured interviews with patients will explain and evaluate the underlying mechanisms of implementing the Mini-AFTERc intervention into routine cancer care from the perspective of breast cancer nurses. Normalisation Process Theory (NPT) will provide a theory-driven framework for addressing this outcome. NPT aims to provide coherence, as well as assessments of cognitive participation, collective action and reflexive monitoring (Murray et al. 2010).
Recruitment rate | Duration of the pilot trial (Approx 2 years)
  Assess number of patients recruited at each site, including those who decline to participate.
Retention rate | Duration of the pilot trial (Approx 2 years)
  Assess number of patients who complete the trial.
Attrition rate | Duration of the pilot trial (Approx 2 years)
  Assess number of patients who do not complete the trial, withdraw or drop-out.
Patient perceived acceptability of the Mini-AFTERc intervention as part of routine cancer care - Determined by theory driven semi-structured interviews | Within 1 month of final follow-up questionnaire
  Semi-structured interviews with patients will explain and evaluate the underlying mechanisms of implementing the Mini-AFTERc intervention into routine cancer care from the perspective of patients. Normalisation Process Theory (NPT) will provide a theory-driven framework for addressing this outcome. NPT aims to provide coherence, as well as assessments of cognitive participation, collective action and reflexive monitoring (Murray et al. 2010).

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Queen Margaret Hospital, Dunfermline, NHS Fife
  - Raigmore Hospital, Inverness, NHS Highlands
  - Western General Hospital, Edinburgh, NHS Lothain
  - Perth Royal Infirmary, Perth, NHS Tayside

REFERENCES:
- [Background] Davidson J, Malloch M, Humphris G. A single-session intervention (the Mini-AFTERc) for fear of cancer recurrence: A feasibility study. Psychooncology. 2018 Nov;27(11):2668-2670. doi: 10.1002/pon.4724. Epub 2018 Apr 30. No abstract available. PMID 29624779
- [Background] Humphris GM, Watson E, Sharpe M, Ozakinci G. Unidimensional scales for fears of cancer recurrence and their psychometric properties: the FCR4 and FCR7. Health Qual Life Outcomes. 2018 Feb 9;16(1):30. doi: 10.1186/s12955-018-0850-x. PMID 29471823
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Mercer SW, Maxwell M, Heaney D, Watt GC. The consultation and relational empathy (CARE) measure: development and preliminary validation and reliability of an empathy-based consultation process measure. Fam Pract. 2004 Dec;21(6):699-705. doi: 10.1093/fampra/cmh621. Epub 2004 Nov 4. PMID 15528286
- [Background] Cruickshank S, Steel E, Fenlon D, Armes J, Scanlon K, Banks E, Humphris G. A feasibility study of the Mini-AFTER telephone intervention for the management of fear of recurrence in breast cancer survivors: a mixed-methods study protocol. Pilot Feasibility Stud. 2017 Jul 20;4:22. doi: 10.1186/s40814-017-0161-8. eCollection 2018. PMID 28748105
- [Background] Humphris G, Ozakinci G. The AFTER intervention: a structured psychological approach to reduce fears of recurrence in patients with head and neck cancer. Br J Health Psychol. 2008 May;13(Pt 2):223-30. doi: 10.1348/135910708X283751. PMID 18492319
- [Background] Bugge C, Williams B, Hagen S, Logan J, Glazener C, Pringle S, Sinclair L. A process for Decision-making after Pilot and feasibility Trials (ADePT): development following a feasibility study of a complex intervention for pelvic organ prolapse. Trials. 2013 Oct 25;14:353. doi: 10.1186/1745-6215-14-353. PMID 24160371
- [Background] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Background] Hartung TJ, Friedrich M, Johansen C, Wittchen HU, Faller H, Koch U, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Weis J, Mehnert A. The Hospital Anxiety and Depression Scale (HADS) and the 9-item Patient Health Questionnaire (PHQ-9) as screening instruments for depression in patients with cancer. Cancer. 2017 Nov 1;123(21):4236-4243. doi: 10.1002/cncr.30846. Epub 2017 Jun 27. PMID 28654189
- [Background] Vodermaier A, Millman RD. Accuracy of the Hospital Anxiety and Depression Scale as a screening tool in cancer patients: a systematic review and meta-analysis. Support Care Cancer. 2011 Dec;19(12):1899-908. doi: 10.1007/s00520-011-1251-4. Epub 2011 Sep 4. PMID 21898134
- [Derived] Brandt NG, McHale CT, Humphris GM. Development and Testing of a Novel Measure to Assess Fidelity of Implementation: Example of the Mini-AFTERc Intervention. Front Psychol. 2020 Nov 25;11:601813. doi: 10.3389/fpsyg.2020.601813. eCollection 2020. PMID 33324299
- [Derived] McHale CT, Cruickshank S, Torrens C, Armes J, Fenlon D, Banks E, Kelsey T, Humphris GM. A controlled pilot trial of a nurse-led intervention (Mini-AFTERc) to manage fear of cancer recurrence in patients affected by breast cancer. Pilot Feasibility Stud. 2020 May 7;6:60. doi: 10.1186/s40814-020-00610-4. eCollection 2020. PMID 32399254